CLINICAL TRIAL: NCT01441453
Title: Value of Transient Elastography in Predicting Postoperative Liver Failure in Patients Undergoing Liver Resection for Hepatocellular Carcinoma.
Brief Title: Transient Elastography in Hepatectomy for Hepatocellular Carcinoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Principal Investigator, Matteo Cescon, MD, PhD, Assistant Professor of Surgery, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FibroBoResect-01
Record Dates: First submitted 2011-09-24; First posted 2011-09-27 (Estimated); Last update posted 2011-09-27 (Estimated); Status verified 2011-09

CONDITIONS: Surgery; Hepatocellular Carcinoma
Keywords: Hepatocellular carcinoma; Cirrhosis; Liver resection; FibroScan
MeSH Terms: conditions — Carcinoma, Hepatocellular; Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Preoperative FibroScan (Other)
  Interventions: Procedure: FibroScan (Transient Elastography measurement)

INTERVENTIONS:
Procedure: FibroScan (Transient Elastography measurement) — Preoperative evaluation of liver stiffness through FibroScan

SUMMARY:
The purpose of this study is to determine whether liver transient elastography performed before the surgical procedure is able to predict liver failure in patients undergoing hepatectomy for hepatocellular carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Patients already scheduled to undergo liver resection fo hepatocellular carcinoma

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)

PRIMARY OUTCOMES:
Cut-off value of liver stiffness measured in kilopascal (kPa) able to predict the occurrence of postoperative liver failure. | Participants will be followed for the duration of postoperative hospital stay, an expected average of 4 weeks
  Definition of the cut-off value in kPa able to predict postoperative liver failure, i.e. the presence of at least one of the following variables: ascites causing a delay in the removal of surgical drainages and/or requiring paracentesis; increase of bilirubin levels >3 mg/dL; alteration of coagulation factors requiring plasma infusion with an INR above 1.50 (with serum bilirubin levels <12mg/dL); renal impairment, defined as blood urea nitrogen >2.00 g/L and/or increase of serum creatinine >2.00 mg/dL requiring only loop diuretics, dopamine/terlipressin, or dialysis.

CONTACTS AND LOCATIONS:
Overall Officials: Matteo Cescon, MD, PhD, Principal Investigator — Policlinico Sant'Orsola-Malpighi, University of Bologna, Italy
Locations (1):
- General Surgery and Organ Transplantation Unit, Policlinico Sant'Orsola-Malpighi, Bologna, Italy